CLINICAL TRIAL: NCT05437926
Title: A Study to Describe the Effectiveness of Arrhythmia Analysis Software for Screening of Sinus Rhythm, Atrial Fibrillation and Premature Beats in Light skin-and Dark Skin Tone Patients
Brief Title: A Study to Describe the Effectiveness of Arrhythmia Analysis Software for Screening of Sinus Rhythm, Atrial Fibrillation and Premature Beats in light-and Dark Skin Tone Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huawei Device Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-2143-WP
Record Dates: First submitted 2022-05-23; First posted 2022-06-29 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Arrhythmia, Cardiac
Keywords: Descriptive study; Arrhythmia analysis software; Cardiac arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Light skin: Light skin Fitzpatrick 1-2 approximately 1/3 with normal sinus rhythm, 1/3 with atrial fibrillation and 1/3 with premature beats
  Interventions: Device: Arrhythmia Analysis Software (software) which runs on a mobile application (Huawei Phone) and uses input from a wearable device (smart watch or smart band).
- Dark skin: Dark skin Fitzpatrick 5-6 approximately 1/3 with normal sinus rhythm, 1/3 with atrial fibrillation and 1/3 with premature beats
  Interventions: Device: Arrhythmia Analysis Software (software) which runs on a mobile application (Huawei Phone) and uses input from a wearable device (smart watch or smart band).

INTERVENTIONS:
Device: Arrhythmia Analysis Software (software) which runs on a mobile application (Huawei Phone) and uses input from a wearable device (smart watch or smart band). — Subjects with or without cardiac arrhythmias and of light skin tone (melanin index <150) or dark skin tone (melanin index >350). Subjects will be divided based on their heart rhythm in three groups: approximately 1/3 with normal sinus rhythm, 1/3 with atrial fibrillation and 1/3 with premature beats

SUMMARY:
The purpose of this study is to describe the Huawei'ssoftware ("Arrhythmia Analysis Software") for the detection of atrial fibrillation, premature beats, and sinus rhythm using photoplethysmography (PPG). Data derived from a wearable device with a PPG sensor (watch or band) in patients with light skin or dark skin tones will be used as an index test. The Huawei software is intended as a pre-screening technology. It should identify candidates who may benefit from further evaluation. The software is not intended to be a diagnostic system.

DETAILED DESCRIPTION:
The purpose of this descriptive study is to describe Huawei's arrhythmia analysis software on PPG data collected with a wearable device (smartwatch or smart band) in people of light and dark skin tones. The study will be conducted at a single research center in The Netherlands. The device under investigation is the Arrhythmia Analysis Software. The Arrhythmia Analysis Software processes a signal from the PPG sensor on a wearable device and displays results data on both the wearable device and mobile phone application.

Data generated from this study will be included in licensing/registration applications for the commercialization of the proposed arrhythmia analysis software. The protocol provides a detailed description of the study and data analysis plan and addresses regulatory requirements relating to ethics approvals, protocol deviations, and disclosure of data. The study will be conducted in compliance with the protocol and all applicable regulatory requirements.

This clinical investigation is a descriptive clinical study at a single research center in which the Huawei Arrhythmia Analysis Software is compared with 12-Lead ECG as the gold standard for arrhythmia detection. Analysis of the ECG output data will be performed by independent physicians who will be blinded to the Arrhythmia Analysis Software output. Also, the physicians deriving data from the Arrhythmia Analysis Software are blinded for analysis of the reference test, the 12-lead ECG. The adjudicated ECG output will then be used to validate the Arrhythmia Analysis Software algorithm.

The 12-lead ECG is the standard for early detection and monitoring of cardiac arrhythmias in Europe and has been used as a comparator.

Prior to enrolling the first patient, the sponsor provides training to the study site personnel to ensure that the study site personnel are fully aware of the research process and are skilled in operating the test instruments.

During the clinical investigation, the investigator must strictly follow the CIP and any related study procedures. The Principal Investigator should perform quality control and supervision to ensure that the investigators strictly follow the study plan. The above measures are implemented throughout the implementation phase of the study to reduce errors or operational errors.

Subjects were screened strictly according to the criteria for selection and exclusion of the CIP to reduce selective bias.

After enrollment, ECG/dynamic ECG results are independently interpreted by ECG physicians with more than 2 years of experience. These physicians were not involved in the ECG collection process and will not be informed of the subject's medical history and past ECG results to reduce the bias of subjective evaluation. Physicians performing the ECG interpretation were blinded to the measurements and outcomes of the Arrhythmia Analysis Software.

Physicians collecting the data from the ECG of the software are blinded for the interpretation of the 12-lead ECG 12-lead ECG was performed at the same time as the ECG from the Arrhythmia Analysis After ECG interpretation has been performed the ECG results were coupled to the Arrhythmia Analysis software output and transferred to the software validation team for analysis.

All the researchers involved in this clinical trial have the relevant working experience to ensure proficiency and standardization of the operation.

An electronic data capture (EDC) system was used to capture the data in this clinical investigation. The system allows for the use of (automated) edit checks and continuous, real-time remote monitoring of trial data by a data manager of the Sponsor. When data issues are detected, the data manager checks and confirms the data by questioning the Investigation Site to avoid recording errors.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 of any sex;
2. Wrist circumference 140 mm - 210 mm;
3. Fitzpatrick skin type 1, 2, 5, or 6 (pre-screening);
4. Melanin Index (MI) <150 or >350 as measured on the inner arm;
5. One of the following conditions, based on past 3 months' history or screening electrocardiogram:

   1. Normal sinus rhythm;
   2. Persistent or permanent or onset atrial fibrillation;
   3. Frequent (>5 beats per minute) premature beats or ongoing premature beats;
6. Willing and able to provide voluntary, written informed consent

Exclusion Criteria:

1. Patients using pacemakers or implantable cardioverter defibrillators (ICDs);
2. Patients with atrioventricular block or bundle branch block;
3. Patients with sinus tachycardia, significant sinus bradycardia, significant sinus arrhythmia, sinus arrest or sick sinus syndrome;
4. Interpositional premature beats, dual-law premature beats, triple-law premature beats, border premature beats or escape beat heart rhythm patients;
5. Patients with atrial tachycardia, atrial flutter, ventricular tachycardia, ventricular flutter or ventricular fibrillation;
6. Patients with a resting heart rate less than 50 times/minute or more than 110 times/minute;
7. Patients with tremor disease or chorea disease that are difficult to cooperate in completing the examination while remaining still;
8. Bullous disease or generalized rash, and other patients not suitable for surface electrode recording;
9. Patients with skin allergies to alcohol;
10. Patients with skin infectious diseases;
11. Patients with a history of mental illness or cognitive impairment;
12. Patients who have participated in other clinical trials that may affect this trial within the past 30 days;
13. Concomitant medication that might interfere with study results;
14. Other situations where the researchers consider it inappropriate for a patient to take part in the trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults >18 years, with or without known heart rhythm irregularities.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-07-21 (Estimated); Study Completion 2023-09-21 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Sinus rhythm | During heart rhythm measurement
  Number of participants with regular sinus P waves (60 to 100 times per minute), P-P distance difference is less than or equal to 0.12s and PR interval > 0.12s
Number of participants with Atrial fibrillation | During heart rhythm measurement
  Number of participants in which the P wave disappears and is replaced by small irregular baseline fluctuations, which vary in shape and amplitude, called f wave; The frequency ranges from 350 to 600 times per minute. The ventricular rate is very irregular, the atrial fibrillation is not treated with drugs, and the atrioventricular conduction is normal, the ventricular rate is usually between 100 and 160 times per minute. The QRS wave morphology is normal. When the ventricular rate is too fast, indoor differential conduction occurs, QRS wave widens and deforms.
Number of participants with Premature atrial beats | During heart rhythm measurement
  Number of participants where the appearance of P-QRS-T is early. Note that there is a difference between P-QRS and sinus P-wave shape, which is the important point in identifying atrial premature beats. Sometimes the P wave is hidden in the T wave of the previous cardiac cycle, causing the T wave to be deformed. The interval between P and R is normal and must be greater than or equal to 0.12s. This means that ectopic excitement comes from the atrium and passes through the atrioventricular node. Sometimes the P-R interval is prolonged, which is caused by the atrioventricular node interference. The QRS waveform of ventricular depolarization after atrial premature beat is similar to that of normal sinus conduction. However, sometimes QRS appears wide deformation, called premature atrial beat with intraventricular differential conduction; Atrial premature beat compensation intervals are many incomplete
Number of participants with Ventricular premature beats | During heart rhythm measurement
  Number of participants which have a QRS wave with broad deformity, time limit ≥ 0.12 s; There are secondary ST-T changes (the direction of T wave is opposite to that of QRS wave) and complete compensation intervals. There was no P wave before and after the QRS wave in the excitation ventricle.
  Agitation reverse conducts agitation at the atrial and produces retrograde P' waves (inverted leads II, III, aVF, upright leads aVR), with three manifestations:
  * (1) retrograde P' wave preceded QRS, P'R interval < 0.12 s;
  * (2) There is no P' wave before and after the QRS wave.
  * (3) Retrograde P' wave after QRS, RP' interval < 0.20 s; VPM with complete/incomplete compensation intervals consult the investigator whether atrial and ventricular premature beats can be combined into one diagnostic criterion.

CONTACTS AND LOCATIONS:
Locations (1):
- Maasstad Hospital, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The results of the research are planned to be shared.